CLINICAL TRIAL: NCT05624632
Title: Cognitive Remote Assessment Using FLAME (CRA-FLAME)
Status: Enrolling by invitation | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CRA- FLAME/BBRC2022
Record Dates: First submitted 2022-11-08; First posted 2022-11-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cognitively unimpaired: Cognitively unimpaired participants from BBRC-sponsored studies
  Interventions: Other: Remote cognitive testing

INTERVENTIONS:
Other: Remote cognitive testing — Remote cognitive testing

SUMMARY:
We aim to use a multimodal approach comprising conventional neuropsychological cognitive tests, fluid and imaging biomarker data, to explore their association with the FLAME unsupervised cognitive computerized assessment. We believe that this would provide critical information to move forward the current research framework in the field.

Participants will be selected from BBRC-sponsored studies, such as the ALFA project (STUDY 45-65 FPM/2012), the ALFA+ cohort study (ALFA - FPM - 0311), the Beta-AARC study (β-AARC_BBRC2020) or the BarcelonaBeta Dementia Prevention Research Clinic study (BBRC-DemPrev-2018)

DETAILED DESCRIPTION:
We aim to use a multimodal approach comprising conventional neuropsychological cognitive tests, fluid and imaging biomarker data, to explore their association with the FLAME unsupervised cognitive computerized assessment. We believe that this would provide critical information to move forward the current research framework in the field.

Participants will be selected from BBRC-sponsored studies, such as the ALFA project (STUDY 45-65 FPM/2012), the ALFA+ cohort study (ALFA - FPM - 0311), the Beta-AARC study (β-AARC_BBRC2020) or the BarcelonaBeta Dementia Prevention Research Clinic study (BBRC-DemPrev-2018)

ELIGIBILITY:
Inclusion Criteria:

Participants must meet ALL the following criteria:

1. To sign the study informed consent form approved by the corresponding authorities.
2. Men and women that have participated/are participating in a BBRC-sponsored study.
3. To accept that:

   * The results obtained in this study may be published in scientific journals and at BBRC's communication channels (e.g. web page)
   * The data gathered may be used in combination with those gathered in other BBRC-sponsored studies in which they may (have) participate(d)

Exclusion Criteria:

1. Not having an ICT literacy enough to access and complete the online tests.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are individuals that have participated/are participating in BBRC-sponsored studies.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
FLAME global composite score | through study completion, an average of 3 years
  calculated by combining information from two web-based online neuropsychological test batteries that are already integrated in a unique platform: the PROTECT Cognitive Tests System (PCTS) (Corbett et al., 2015) and the CogTrackTM (Wesnes et al., 2017)

CONTACTS AND LOCATIONS:
Locations (1):
- BarcelonaBeta Brain Research Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No